CLINICAL TRIAL: NCT03463213
Title: She's Healthy and Empowered (SHE Tribe): A Social Networked-based Peer-facilitated Intervention to Improve Health Behavior Among Women in Underserved Communities
Brief Title: SHE Tribe: An Intervention to Improve Health Behavior Among Women in Underserved Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: YMCA of Metropolitan Fort Worth (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Emily Spence-Almaguer, Associate Dean; Associate Professor, University of North Texas Health Science Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-148; U54MD006882-06 (NIH)
Record Dates: First submitted 2018-02-10; First posted 2018-03-13 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Health Promotion
Keywords: health behavior; chronic disease prevention; healthy lifestyle
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a feasibility study with a single group pre/post outcome design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHE Tribe (Experimental): SHE Tribe is a social network-based peer-facilitated intervention to promote adoption of health behaviors
  Interventions: Behavioral: SHE Tribe

INTERVENTIONS:
Behavioral: SHE Tribe — Social network-based peer-facilitated intervention to promote adoption of health behavior

SUMMARY:
While healthy lifestyle behaviors have been identified as instrumental to preventing chronic disease, programs to successfully promote healthy behavior adoption in underserved communities have had limited sustainable success. SHE Tribe is a culturally tailored, social network intervention created through CBPR to overcome previously identified barriers and improve health behavior among women in underserved communities.

DETAILED DESCRIPTION:
The leading causes of death for women in the United States are heart disease, cancer, and stroke. Chronic diseases disproportionately affect underserved communities where race, poverty, education-level, healthcare access, and other social and environmental determinants intersect. African-American (AA) and Hispanic women are at particularly high risk for diabetes-related mortality 1 and are more likely than white women to be functionally impacted by chronic disease . Factors associated with increased disease risk include physical inactivity, poor nutrition, obesity, underutilization of health screenings, and high stress/allostatic load . While healthy lifestyle behaviors have been identified as instrumental to preventing chronic disease, programs to successfully promote healthy behavior adoption in underserved communities have had limited sustainable success, due in part to perceived relevance of program outcomes, lack of cultural tailoring, access to care, and lack of social support for health behavior change.

The Texas Center for Health Disparities received National Institute of Minority Health and Health Disparities funding to address women's chronic health conditions through community outreach and research strategies from 2012-2017. A workgroup of community members, former research and program participants, and University of North Texas Health Science Center faculty and staff utilized a Community-Based Participatory Research (CBPR) process to design SHE Tribe (She's Healthy and Empowered), a social-network based initiative to support healthy behavior adoption among women in underserved communities. This effort was based on earlier findings that women in underserved neighborhoods were often resistant to participating in a "disease-labeled" intervention (e.g., obesity prevention) and expressed a desire to practice wellness-oriented behaviors that have been adapted for their social and cultural groups. These findings were consistent with the growing body of literature indicating that being "healthy and strong" is perceived as more desirable than engaging in a program where the explicit expectation is to lose weight. As part of the development process, the workgroup sought to develop a sustainable, evidence-based approach that would appeal to underserved communities that are disproportionately impacted by chronic disease.

Components of SHE Tribe include evidence-based characteristics associated with the adoption and maintenance of health behaviors: a) incorporating social network to promote healthy activities, b) setting goals that are specific to the needs and interests of the individual , c) self-monitoring of desired behaviors, d) motivational interviewing-based dialogue that promotes intrinsic motivation to change, e) choosing small units of change for the purpose of habit formation, and f) combining practice and reflection to promote integration with existing life patterns and beliefs. The advantage of SHE Tribe over previous models is its explicit use of social networks and reliance on a broader set of activities that are consistent with a healthy lifestyle rather than disease. SHE Tribe was initially pilot-tested with a small cohort of 5 peer facilitators. Based on their feedback, it was then enhanced to include telephone or tablet-based assessment and tailored feedback at the beginning (baseline) and end of each 5-session cycle. The current version is being pilot-tested as a community-initiated project, and as such includes only a basic set of assessment tools that are necessary to make the intervention work. The purpose of this 2-year exploratory submission is to examine the effects of SHE Tribe on key health outcomes such as health self-management, coping, diet, activity, and social network health norms.

AIM 1. Determine whether SHE Tribe can be feasibly implemented with groups of women from communities at high risk for chronic health conditions. The research team will examine the characteristics of women recruited to SHE Tribe to determine whether the network-based recruitment is an effective method for reaching the underserved communities. This will include a review of audio-recorded sessions, session summary reports, and semi-structured interviews with participants and facilitators to understand the perceived value and adoption of different intervention components.

AIM 2. Examine how health behaviors are adopted by individuals and diffused through social networks. At the individual level: Using validated measures, the research team determine which goals are selected and the relationship between goal selection, key health outcomes, and activation of health behavior self-management. At the interpersonal level: Using a social network analysis instrument which measures participants' perceptions of identified individuals in their networks, the research team will examine the diffusion of healthy lifestyle norms.

The impact of this study will be the refinement of an intervention that supports sustainability and reach in underserved communities that are at high-risk for chronic diseases. The emphasis on a constellation of healthy behaviors and the use of peer facilitators will appeal to the cultural identities of women residing in underserved and/or high poverty communities.

ELIGIBILITY:
Inclusion Criteria:

* Female
* representative of underserved community (determined by race, ethnicity, socioeconomic status, and/or neighborhood)
* 18 and older

Exclusion Criteria:

* Males
* Children

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must self-represent as a female
Enrollment: 240 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Habits Tracking | Baseline and 8 weeks.
  This tool includes 42 items representing tracking and monitoring behaviors, such as weighing oneself, keeping a food diary, etc... Each is answered with a yes/no (0/1) response. Scores range from 0 to 42. The questionnaire is administered at baseline and again at 8 weeks. The desired outcome is an increase in the total score between baseline and 8 weeks.

SECONDARY OUTCOMES:
Social Support for Diet and Physical Activity | Baseline and 8 weeks.
  These 11 items are adapted from the Patient Assessment and Counseling for Exercise (PACE+ Women: Measurement Questionnaire). Scores range from 11 to 44, with higher scores indicating a greater social support for healthy lifestyle choices associated with diet and exercise.
Coping with stress | Baseline and 8 weeks.
  These 10 questions include 5 subscales from the Brief COPE tool which measure use of emotional support, use of instrumental support, positive reframing, planning and religion. Each sub-scale score ranges from 0 to 4 with higher values reflecting better coping strategies.
Body Appreciation Scale (BAS-2) | Baseline and 8 weeks.
  This is a 10 item scale measuring body positivity. Scores are based on mean values of all items.
Healthy Lifestyle Activation | Baseline and 8 weeks.
  This tool includes 7 items that measure health-related efficacy, agency, and self-management. Each item is ranked on a scale of 1 to 10 with overall scores ranging from 7 to 70.
Fruit and vegetable consumption | Baseline and 8 weeks.
  This item is from the Patient Assessment and Counseling for Exercise (PACE+ Women: Measurement Questionnaire) and measures self-reported days of purposeful physical activity (30 minutes or more) during a typical week. Scores range from 0 to 7 with higher values reflecting more frequent physical activity.
Physical activity days | Baseline and 8 weeks.
  This item is from the Patient Assessment and Counseling for Exercise (PACE+ Women: Measurement Questionnaire) and measures self-reported daily consumption of fruit and vegetables servings.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Spence-Almaguer, PhD, Principal Investigator — UNT Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sudano JJ, Baker DW. Explaining US racial/ethnic disparities in health declines and mortality in late middle age: the roles of socioeconomic status, health behaviors, and health insurance. Soc Sci Med. 2006 Feb;62(4):909-22. doi: 10.1016/j.socscimed.2005.06.041. Epub 2005 Aug 2. PMID 16055252
- [Background] Lantz PM, House JS, Lepkowski JM, Williams DR, Mero RP, Chen J. Socioeconomic factors, health behaviors, and mortality: results from a nationally representative prospective study of US adults. JAMA. 1998 Jun 3;279(21):1703-8. doi: 10.1001/jama.279.21.1703. PMID 9624022
- [Background] Kington RS, Smith JP. Socioeconomic status and racial and ethnic differences in functional status associated with chronic diseases. Am J Public Health. 1997 May;87(5):805-10. doi: 10.2105/ajph.87.5.805. PMID 9184510
- [Background] Mosca L. Guidelines for prevention of cardiovascular disease in women: a summary of recommendations. Prev Cardiol. 2007 Fall;10 Suppl 4:19-25. doi: 10.1111/j.1520-037x.2007.07255.x. PMID 17917527
- [Background] Geronimus AT, Hicken M, Keene D, Bound J. "Weathering" and age patterns of allostatic load scores among blacks and whites in the United States. Am J Public Health. 2006 May;96(5):826-33. doi: 10.2105/AJPH.2004.060749. Epub 2005 Dec 27. PMID 16380565
- [Background] Bauer UE, Briss PA, Goodman RA, Bowman BA. Prevention of chronic disease in the 21st century: elimination of the leading preventable causes of premature death and disability in the USA. Lancet. 2014 Jul 5;384(9937):45-52. doi: 10.1016/S0140-6736(14)60648-6. Epub 2014 Jul 1. PMID 24996589
- [Background] Nelson D, Harris A, Horner-Ibler B, Harris KS, Burns E. Hearing the Community: Evolution of a Nutrition and Physical Activity Program for African American Women to Improve Weight. J Health Care Poor Underserved. 2016;27(2):560-7. doi: 10.1353/hpu.2016.0088. PMID 27180695
- [Background] Bacon L, Aphramor L. Weight science: evaluating the evidence for a paradigm shift. Nutr J. 2011 Jan 24;10:9. doi: 10.1186/1475-2891-10-9. PMID 21261939
- [Background] Bacon L, Keim NL, Van Loan MD, Derricote M, Gale B, Kazaks A, Stern JS. Evaluating a 'non-diet' wellness intervention for improvement of metabolic fitness, psychological well-being and eating and activity behaviors. Int J Obes Relat Metab Disord. 2002 Jun;26(6):854-65. doi: 10.1038/sj.ijo.0802012. PMID 12037657
- [Background] Kumanyika SK, Wadden TA, Shults J, Fassbender JE, Brown SD, Bowman MA, Brake V, West W, Frazier J, Whitt-Glover MC, Kallan MJ, Desnouee E, Wu X. Trial of family and friend support for weight loss in African American adults. Arch Intern Med. 2009 Oct 26;169(19):1795-804. doi: 10.1001/archinternmed.2009.337. PMID 19858438
- [Background] Anderson JW, Konz EC, Frederich RC, Wood CL. Long-term weight-loss maintenance: a meta-analysis of US studies. Am J Clin Nutr. 2001 Nov;74(5):579-84. doi: 10.1093/ajcn/74.5.579. PMID 11684524
- [Background] Fitzgibbon ML, Tussing-Humphreys LM, Porter JS, Martin IK, Odoms-Young A, Sharp LK. Weight loss and African-American women: a systematic review of the behavioural weight loss intervention literature. Obes Rev. 2012 Mar;13(3):193-213. doi: 10.1111/j.1467-789X.2011.00945.x. Epub 2011 Nov 10. PMID 22074195
- [Background] Warsi A, Wang PS, LaValley MP, Avorn J, Solomon DH. Self-management education programs in chronic disease: a systematic review and methodological critique of the literature. Arch Intern Med. 2004 Aug 9-23;164(15):1641-9. doi: 10.1001/archinte.164.15.1641. PMID 15302634
- [Background] Samuel-Hodge CD, Johnson CM, Braxton DF, Lackey M. Effectiveness of Diabetes Prevention Program translations among African Americans. Obes Rev. 2014 Oct;15 Suppl 4:107-24. doi: 10.1111/obr.12211. PMID 25196409
- [Background] Brady TJ, Murphy L, O'Colmain BJ, Beauchesne D, Daniels B, Greenberg M, House M, Chervin D. A meta-analysis of health status, health behaviors, and health care utilization outcomes of the Chronic Disease Self-Management Program. Prev Chronic Dis. 2013;10:120112. doi: 10.5888/pcd10.120112. PMID 23327828
- [Background] Yancey AK, Ortega AN, Kumanyika SK. Effective recruitment and retention of minority research participants. Annu Rev Public Health. 2006;27:1-28. doi: 10.1146/annurev.publhealth.27.021405.102113. PMID 16533107
- [Background] Chin MH, Clarke AR, Nocon RS, Casey AA, Goddu AP, Keesecker NM, Cook SC. A roadmap and best practices for organizations to reduce racial and ethnic disparities in health care. J Gen Intern Med. 2012 Aug;27(8):992-1000. doi: 10.1007/s11606-012-2082-9. PMID 22798211
- [Background] Hibbard JH, Greene J, Becker ER, Roblin D, Painter MW, Perez DJ, Burbank-Schmitt E, Tusler M. Racial/ethnic disparities and consumer activation in health. Health Aff (Millwood). 2008 Sep-Oct;27(5):1442-53. doi: 10.1377/hlthaff.27.5.1442. PMID 18780935
- [Background] Green LW, Ottoson JM, Garcia C, Hiatt RA. Diffusion theory and knowledge dissemination, utilization, and integration in public health. Annu Rev Public Health. 2009;30:151-74. doi: 10.1146/annurev.publhealth.031308.100049. PMID 19705558
- [Background] Pearson ES. Goal setting as a health behavior change strategy in overweight and obese adults: a systematic literature review examining intervention components. Patient Educ Couns. 2012 Apr;87(1):32-42. doi: 10.1016/j.pec.2011.07.018. Epub 2011 Aug 17. PMID 21852063
- [Background] Rubak S, Sandbaek A, Lauritzen T, Christensen B. Motivational interviewing: a systematic review and meta-analysis. Br J Gen Pract. 2005 Apr;55(513):305-12. PMID 15826439
- [Background] Burke LE, Wang J, Sevick MA. Self-monitoring in weight loss: a systematic review of the literature. J Am Diet Assoc. 2011 Jan;111(1):92-102. doi: 10.1016/j.jada.2010.10.008. PMID 21185970
- [Background] Hill JO. Can a small-changes approach help address the obesity epidemic? A report of the Joint Task Force of the American Society for Nutrition, Institute of Food Technologists, and International Food Information Council. Am J Clin Nutr. 2009 Feb;89(2):477-84. doi: 10.3945/ajcn.2008.26566. Epub 2008 Dec 16. PMID 19088151
- [Background] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Background] Harmon BE, Forthofer M, Bantum EO, Nigg CR. Perceived influence and college students' diet and physical activity behaviors: an examination of ego-centric social networks. BMC Public Health. 2016 Jun 6;16:473. doi: 10.1186/s12889-016-3166-y. PMID 27267371
- [Background] Latkin CA, Knowlton AR. Social Network Assessments and Interventions for Health Behavior Change: A Critical Review. Behav Med. 2015;41(3):90-7. doi: 10.1080/08964289.2015.1034645. PMID 26332926
- [Background] Michie S, Abraham C, Whittington C, McAteer J, Gupta S. Effective techniques in healthy eating and physical activity interventions: a meta-regression. Health Psychol. 2009 Nov;28(6):690-701. doi: 10.1037/a0016136. PMID 19916637
- [Background] Stevanovic D. Quality of Life Enjoyment and Satisfaction Questionnaire-short form for quality of life assessments in clinical practice: a psychometric study. J Psychiatr Ment Health Nurs. 2011 Oct;18(8):744-50. doi: 10.1111/j.1365-2850.2011.01735.x. Epub 2011 May 5. PMID 21896118
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Greene J, Hibbard JH. Why does patient activation matter? An examination of the relationships between patient activation and health-related outcomes. J Gen Intern Med. 2012 May;27(5):520-6. doi: 10.1007/s11606-011-1931-2. PMID 22127797
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Beaudreau SA, Spira AP, Stewart A, Kezirian EJ, Lui LY, Ensrud K, Redline S, Ancoli-Israel S, Stone KL; Study of Osteoporotic Fractures. Validation of the Pittsburgh Sleep Quality Index and the Epworth Sleepiness Scale in older black and white women. Sleep Med. 2012 Jan;13(1):36-42. doi: 10.1016/j.sleep.2011.04.005. Epub 2011 Oct 26. PMID 22033120
- [Background] Carlson JA, Sallis JF, Wagner N, Calfas KJ, Patrick K, Groesz LM, Norman GJ. Brief physical activity-related psychosocial measures: reliability and construct validity. J Phys Act Health. 2012 Nov;9(8):1178-86. doi: 10.1123/jpah.9.8.1178. Epub 2011 Dec 27. PMID 22207589
- [Background] Miura S, Yamaguchi Y, Urata H, Himeshima Y, Otsuka N, Tomita S, Yamatsu K, Nishida S, Saku K. Efficacy of a multicomponent program (patient-centered assessment and counseling for exercise plus nutrition [PACE+ Japan]) for lifestyle modification in patients with essential hypertension. Hypertens Res. 2004 Nov;27(11):859-64. doi: 10.1291/hypres.27.859. PMID 15824468
- [Background] Calfas KJ, Sallis JF, Zabinski MF, Wilfley DE, Rupp J, Prochaska JJ, Thompson S, Pratt M, Patrick K. Preliminary evaluation of a multicomponent program for nutrition and physical activity change in primary care: PACE+ for adults. Prev Med. 2002 Feb;34(2):153-61. doi: 10.1006/pmed.2001.0964. PMID 11817910
- See also: Diabetes Prevention Programs: Effectiveness and Value — http://www.icer-review.org